CLINICAL TRIAL: NCT05501756
Title: Precision Alemtuzumab Dosing for Allogeneic Hematopoietic Cell Transplantation in Non-Malignant Diseases
Brief Title: Precision Alemtuzumab Dosing for Allogeneic Hematopoietic Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0447
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Allogeneic Hematopoietic Cell Transplantation
MeSH Terms: interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Alemtuzumab (Experimental): Patients will be given 10 mg/m2 alemtuzumab divided over days -14, -13, and -12. The first dose should be limited to no more than 3 mg per the manufacturer's recommendation. If the calculated daily dose is greater than 3 mg, the first dose (day -14) should be limited to 3 mg and the remainder of the dosing should be divided over days -13 and -12.
  Alemtuzumab will be drawn into a sterile syringe and given to patients subcutaneously.
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab (Campath®) is a recombinant DNA-derived humanized monoclonal antibody directed against CD52. Alemtuzumab is produced in mammalian cell (Chinese hamster ovary) suspension culture in a medium containing neomycin. Neomycin is not detectable in the final product. Alemtuzumab is a sterile, clear, colorless, isotonic pH 6.8-7.4 solution for injection. Alemtuzumab is supplied in single-use clear glass ampules containing 30 mg of Alemtuzumab in 3 mL of solution. A single use vial of alemtuzumab contains 30 mg alemtuzumab, 8 mg sodium chloride, 1.44 mg dibasic sodium phosphate, 0.2 mg potassium chloride, 0.2 mg monobasic potassium phosphate, 0.1 mg polysorbate 80, and 0.0187 mg disodium edetate dihydrate.
  Other Names: Campath

SUMMARY:
Alemtuzumab is an antibody that reduces the strength of the immune system that is given in preparation for allogeneic hematopoietic cell transplant (HCT). In this research study the investigators want to find out if they can adjust the dose of alemtuzumab used as part of allogeneic HCT to target the level of Day 0 (the planned day of graft infusion) to an optimal therapeutic window of 0.15-0.9 ug/mL.

DETAILED DESCRIPTION:
Alemtuzumab levels at Day 0 can affect:

* the chances of developing acute graft versus host disease (GVHD), which is an immune reaction of the donor cells against your own tissues
* the chances of developing mixed chimerism, which is having a mixture of your own cells and donor cells after HCT, and
* recovery of your immune system following transplant.

High levels of alemtuzumab are associated with more mixed chimerism and slower immune recovery, while low levels are associated with more acute GVHD. The investigators have developed a plan to adjust the alemtuzumab dose for patients to target Day 0 levels to fall within an ideal effective range of 0.15-0.9 ug/mL. This range may minimize the risks of these complications. The investigators are conducting this study to determine if the current plan for alemtuzumab dosing will be successful in the majority of patients and evaluate the impact on the clinical outcomes of acute GVHD, mixed chimerism, and immune recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing allogeneic HCT at CCHMC with an alemtuzumab-containing preparative regimen for treatment of a non-malignant disease are eligible.
* For the first 7 patients, patients must have a 10/10 HLA matched related or unrelated stem cell donor, or be receiving a CD34+ selected stem cell product. After the first 7 patients, any donor match may be allowed after data review by the BMT clinicians and the PI.

Exclusion Criteria:

* Patients with a history of anaphylaxis to alemtuzumab.
* Patients who have previously received alemtuzumab and have not cleared alemtuzumab prior to the start of the preparative regimen.
* Life expectancy less than 4 weeks.
* Patients receiving dialysis or plasmapheresis at the time of the start of the conditioning regimen.
* Failure to sign informed consent and/or assent, or inability to undergo informed consent process.
* It is not medically advisable to obtain the specimens necessary for this study.
* Not able to tolerate subcutaneous dosing (patients with severe skin conditions).
* Patients with cancer.
* Patients whose clinical condition suggest there may be inability to successfully perform the PK modeling such as, but not limited to, active flaring of hemophagocytic lymphohistiocytosis in which excessive lymphoproliferation may significantly alter the target-mediated clearance of alemtuzumab and prevent observation of non-target mediated clearance which is needed for robust modeling.
* Patients whose pre-alemtuzumab level reveals an interfering substance which prevents accurate measurement of alemtuzumab.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Alemtuzumab levels | 100 days
  Number of patients who have alemtuzumab levels in the optimal therapeutic range on Day 0.

SECONDARY OUTCOMES:
CD4+ T cell count | 100 days
  CD4+ T cell count in patients who achieve the target window compared to patients who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Parinda Mehta, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No